CLINICAL TRIAL: NCT02085577
Title: The Effect of Intraoperative Ketamine on Opioid Consumption and Pain After Spine Surgery in Opioid-dependent Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Rikke Vibeke Nielsen, MD, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM3-RS-2014; 2014-000839-16 (EudraCT Number)
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Postoperative Pain; Chronic Pain; Analgesics
Keywords: Morphine consumption; Postoperative pain; Ketamine; Side effects; Spine surgery; Chronic pain
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Ketamine; Sodium Chloride; Acetaminophen; Morphine; Ondansetron; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): * (S)-(+)-Ketamine Hydrochloride Solution 25 mg/ml bolus 0.5 mg/kg administered immediately after induction of anesthesia, followed by infusion ketamine 0,25 mg/kg/h terminated at last suture to the skin.
  * Morphine. Morphine Sulphate 1 mg/ml, bolus 0.4 mg/kg administered 45 min before expected awakening.
  * Escape sufentanil. Sufentanil 5 microgram/ml, bolus 5 micrograms administered by the anaesthetic nurse in the operating room if the patient is in pain upon awakening.
  * Morphine. PCA-morphine, bolus 2.5 mg, lock-out-time 5 min. Concentration : Morphine sulphate 1 mg/ml.
  * Escape morphine. Morphine Sulphate 1 mg/ml, bolus 2.5 mg administered by the PACU nurse on request of the patient for the first hour postoperatively.
  * Ondansetron 2 mg/ml, 4 mg iv in case of moderate to severe nausea, supplemented by 1 mg iv if needed
  * Paracetamol 1 g orally 1 h preoperatively and every 6 h after extubation time during the first 24 h.
  * The patients usual daily opioids
  Interventions: Drug: (S)-(+)-Ketamine Hydrochloride Solution 25 mg/ml; Drug: Paracetamol 1 g; Drug: Morphine Sulphate 1 mg/ml; Drug: Ondansetron 2 mg/ml; Drug: Usual daily opioids; Drug: Sufentanil 5 microgram/ml
- Placebo (Placebo Comparator): * Isotonic sodium chloride 0.9 percent 0.02 ml/kg administered immediately after induction of anesthesia, followed by infusion isotonic sodium chloride 0.01 ml/kg/h terminated at last suture to the skin.
  * Morphine. Morphine Sulphate 1 mg/ml, bolus 0.4 mg/kg administered 45 min before expected awakening.
  * Escape sufentanil. Sufentanil 5 microgram/ml, bolus 5 micrograms administered by the anaesthetic nurse in the operating room if the patient is in pain upon awakening.
  * Morphine. PCA-morphine, bolus 2.5 mg, lock-out-time 5 min. Concentration : Morphine sulphate 1 mg/ml.
  * Escape morphine. Morphine Sulphate 1 mg/ml, bolus 2.5 mg administered by the PACU nurse on request of the patient for the first hour postoperatively.
  * Ondansetron 2 mg/ml, 4 mg iv in case of moderate to severe nausea, supplemented by 1 mg iv if needed
  * Paracetamol 1 g orally 1 h preoperatively and every 6 h after extubation time during the first 24 h.
  * The patients usual daily opioids
  Interventions: Drug: Isotonic sodium chloride 0.9 percent; Drug: Paracetamol 1 g; Drug: Morphine Sulphate 1 mg/ml; Drug: Ondansetron 2 mg/ml; Drug: Usual daily opioids; Drug: Sufentanil 5 microgram/ml

INTERVENTIONS:
Drug: (S)-(+)-Ketamine Hydrochloride Solution 25 mg/ml — Ketamine (25 mg/ml) bolus 0.5 mg/kg administered immediately after induction of anesthesia, followed by infusion ketamine 0,25 mg/kg/hour that is terminated when the last suture to the skin has been performed.
  Other Names: Ketamine
  Arms: Ketamine
Drug: Isotonic sodium chloride 0.9 percent — Isotonic sodium chloride 0.9 percent 0.02 ml/kg administered immediately after induction of anesthesia, followed by infusion isotonic sodium chloride 0.01 ml/kg/hour that is terminated when the last suture to the skin has been performed.
  Other Names: Isotonic saline
  Arms: Placebo
Drug: Paracetamol 1 g — Paracetamol 1 g orally 1 hour preoperatively and every 6 hours after extubation time during the first 24 hours.
  Other Names: Paracetamol
Drug: Morphine Sulphate 1 mg/ml — Morphine Sulphate 1 mg/ml administered as patient-controlled analgesia (PCA, bolus 2.5 mg, lockout 5 minutes) 0-24 hours postoperatively
  Other Names: Morphine
Drug: Morphine Sulphate 1 mg/ml — Morphine Sulphate 1 mg/ml, bolus 2.5 mg administered by the PACU nurse on request of the patient for the first hour postoperatively.
  Other Names: Morphine
Drug: Ondansetron 2 mg/ml — Ondansetron 2 mg/ml 4 mg iv in case of moderate to severe nausea, supplemented by Ondansetron 1 mg iv if needed
  Other Names: Zofran
Drug: Usual daily opioids — The patients usual daily opioid consumption are administered during the study period
  Other Names: Morphine
Drug: Morphine Sulphate 1 mg/ml — Morphine Sulphate 1 mg/ml, bolus 0.4 mg/kg administered 45 minutes before expected awakening.
  Other Names: Morphine
Drug: Sufentanil 5 microgram/ml — Sufentanil 5 microgram/ml, bolus 5 micrograms administered by the anaesthetic nurse in the operating room if the patient is in pain upon awakening.
  Other Names: Sufentanil

SUMMARY:
Patients with a daily use of opioids may develop higher postoperative pain levels, often need high doses of morphine and therefore their pain may be difficult to treat. A low dose of an old anesthetic drug, ketamine, administered during surgery can possibly reduce pain and morphine consumption in these patients. Our purpose is to investigate the effect of low dose ketamine on morphine consumption and pain after spine surgery in patients with a daily use of opioids. Our hypothesis is that low dose ketamine can reduce morphine consumption, pain and side-effects after spine surgery.

DETAILED DESCRIPTION:
Opioid-dependent patients can develop hyperalgesia and often have a high opioid consumption postoperatively due to opioid tolerance. Intraoperative ketamine in subanesthetic doses can possibly reduce hyperalgesia and reduce opioid-tolerance in these patients. Ketamine is a non-competitive N-methyl-D-aspartate (NMDA) receptor antagonist that works by blocking the NMDA receptors in the central and peripheral nerve system. It can be used for general anesthesia but the drug also has other properties including lowering of central excitability and reducing postoperative opioid tolerance by modeling the opioid receptors. Further more it can possibly reduce chronic pain by blocking wind-up effect when blocking the NMDA receptors.

Our purpose is to investigate the effect of intraoperative ketamine on opioid consumption and pain after spine surgery in opioid-dependent patients. Our hypothesis is that ketamine can reduce opioid consumption and reduce postoperative pain and side effects compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lumbar spinal fusion surgery in general anesthesia.
* Daily use of opioids for a minimum of 6 weeks preoperatively (morphine, ketobemidone, oxycodone, fentanyl, tramadol and/or buprenorphine).
* Back pain for a minimum of 3 months preoperatively.
* Age > 18 years and < 85 years.
* ASA 1-3.
* BMI > 18 and < 40.
* Fertile women need to have a negative urine HCG pregnancy test.
* Patients who have given their written informed consent to participate in the study after understanding the content and limitations of the study

Exclusion Criteria:

* Participation in another concomitant drug trial.
* Patients who do not understand or speak Danish.
* Allergy to the drugs used in the trial.
* Abuse of drugs - as assessed by the investigator.
* Daily methadone use.
* Increased intraocular pressure - assessed from the patients chart.
* Uncontrolled hypertension - assessed from the patients chart.
* Previous and current psychotic episodes - assessed from the patients chart

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 0-24 hours postoperatively
  Total intravenous morphine consumption, other than the patients usual opioid use, 0- 24 hours postoperatively, administered as patient-controlled analgesia ((PCA), bolus 2.5 mg, lockout 5 minutes)

SECONDARY OUTCOMES:
Pain during mobilization | 2, 6, 12, 18 and 24 hours postoperatively
  Pain score during active mobilization, measured on a visual analogue scale (VAS) (0-100 mm), defined as a standardized movement from recumbent position to sitting on the bedside at 2, 6, 12, 18 and 24 hours postoperatively, the worst pain from the movement is registered. The endpoint, VAS-mobilization, will be calculated as area under the curve (AUC) (2-24h) from these measurements.
Pain at rest | 2, 6, 12, 18 & 24 hours postoperatively
  Pain score at rest, measured on a visual analogue scale (VAS) (0-100 mm), at 2, 6, 12, 18 and 24 hours postoperatively. The endpoint, VAS-rest, will be calculated as area under the curve (AUC) (2-24h) from these measurements.
Nausea | 2, 6, 12, 18 & 24 hours postoperatively
  Level of nausea (none, mild, moderate, severe) (0-24h), measured at 2, 6, 12, 18 and 24 hours postoperatively.
Vomiting | 0-2, 2-6, 6-12, 12-18, 18-24 hours postoperatively
  Number of vomiting episodes (0-24 hours), registered in the periods 0-2, 2-6, 6-12, 12-18, 18-24 hours postoperatively.
Ondansetron | 0-24 hours postoperatively
  Consumption of ondansetron (mg) during 0-24 hours postoperatively.
Sedation | 2, 6, 12, 18 & 24 hours postoperatively
  Level of sedation (none, mild, moderate, severe) (0-24 h) registered at time 2, 6, 12, 18 and 24 hours postoperatively.
Hallucinations and nightmares | 0-24 hours postoperatively
  Episodes of hallucinations and nightmares (yes/no) in the period 0-24 hours postoperatively.
Chronic pain | 6 months postoperatively
  Level of chronic pain and daily use of opioids assessed by the validated questionnaires EQ50, OWESTRY and DN4 at 6 months postoperatively.
Chronic pain | 12 months postoperatively
  Level of chronic pain and daily use of opioids assessed by the validated questionnaires EQ50, OWESTRY and DN4 at 12 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Rikke V Nielsen, MD, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Department of Anaesthesiology, Glostrup Hospital, Glostrup Municipality, Denmark

REFERENCES:
- [Background] Loftus RW, Yeager MP, Clark JA, Brown JR, Abdu WA, Sengupta DK, Beach ML. Intraoperative ketamine reduces perioperative opiate consumption in opiate-dependent patients with chronic back pain undergoing back surgery. Anesthesiology. 2010 Sep;113(3):639-46. doi: 10.1097/ALN.0b013e3181e90914. PMID 20693876